CLINICAL TRIAL: NCT04398966
Title: Prostatic Artery Embolization vs Medication for Benign Prostatic Hyperplasia: Single Subject Study Design
Brief Title: Prostatic Artery Embolization vs Medication for Benign Prostatic Hyperplasia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The principal investigator is leaving UNC and there is no other faculty to continue the research study.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Terumo Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-0472
Record Dates: First submitted 2020-05-18; First posted 2020-05-22 (Actual); Results first posted 2024-04-03 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2023-10

CONDITIONS: BPH; Enlarged Prostate (BPH); Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- PAE Procedure (Experimental): This will be a single arm, uncontrolled, non-blinded study of PAE using HydroPearl Beads in a small population of 30 subjects with benign prostate hyperplasia (BPH)
  Interventions: Device: Prostatic Artery Embolization (HydroPearl® compressible microspheres)

INTERVENTIONS:
Device: Prostatic Artery Embolization (HydroPearl® compressible microspheres) — Embolic material
  Other Names: HydroPearl® compressible microspheres (75 to 400 µm)

SUMMARY:
Purpose: The purpose of this study is to determine if prostatic artery embolization (PAE) is as effective as medication (non-inferiority) in reducing urinary symptoms due to benign prostatic hyperplasia (BPH) and to determine if PAE will result in less adverse events compared to medication in individual patients.

Participants: Study subjects will be 30 men who have taken BPH medication for at least 6 months and planning to undergo PAE. Subjects will be enrolled across 3 sites.

Procedures (methods): This will be a single arm, non-blinded study of PAE using HydroPearl Beads. Subjects will be compared to themselves. The study will involve 6 study visits: an enrollment/baseline visit, the PAE procedure, and 1 day, 3 month, 6 month, and 12 month follow-up visits. Subjects will complete questionnaires and uroflowmetry testing at baseline and each follow-up visit. Subjects will also obtain an MRI at baseline and their 6 month follow-up visit.

DETAILED DESCRIPTION:
This will be a single arm, uncontrolled, non-blinded study of PAE using HydroPearl Beads in a small population of 30 subjects with benign prostate hyperplasia (BPH) to investigate the effectiveness of prostatic artery embolization (PAE) relative to previous medication alone for reducing urinary symptoms due to BPH. Secondary aims will be to assess adverse effects of medication vs adverse events secondary to PAE as well as Quality of Life scores on medication vs after PAE.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age ≥ 40
* Prostate gland measures ≥50 grams measured by MRI, CT, or ultrasound
* Have previously taken BPH medications including either alpha blockers, 5-alpha reductase inhibitors or the combination of both for 6 months
* Capable of giving informed consent
* Life expectancy greater than 1 year

Exclusion Criteria:

* Severe vascular disease as defined by severe arterial calcification seen on prior imaging, history of lower extremity or pelvic bypass grafts or history of lower extremity or pelvic arterial stenting. For patients that do not have prior imaging at UNC, we will rule out suspected severe arterial calcification given their medical history.
* Uncontrolled diabetes mellitus which is defined as Hemoglobin A1C >8%
* Patients currently taking SGLT2 inhibitors (cana-, dapa-, empa-, and ertu- gliflozin) due to their diuretic effects
* A smoking history of 20 pack-year or greater obtained by patient report
* Prior myocardial infarction
* A stroke within the last 6 months
* Unstable angina
* Immunosuppression
* Neurogenic bladder and/or sphincter abnormalities secondary to Parkinson's disease, multiple sclerosis, cerebral vascular accident, diabetes, etc.
* Complete urinary retention
* Impaired kidney function (serum creatinine level > 1.8 mg/dl or a glomerular filtration rate < 60 as approximated using serum creatinine levels) unless anuric and on dialysis.
* Confirmed or suspected bladder cancer as assessed based on patients' medical history or current hematuria
* Urethral strictures, bladder neck contracture, or other potentially confounding bladder pathology
* Ongoing urogenital infection. For patients with symptoms of a urogenital infection (dysuria, fever, etc.), a urinalysis will be obtained.
* Previous pelvic radiation or radical pelvic surgery
* Confirmed malignancy of the prostate or a history of prostate cancer
* Contrast hypersensitivity refractory to standard medications (antihistamines, steroids)

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyeon Yu, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: 9 to 36 months following publication
Access Criteria: The investigator who proposes to use the data has approval from an IRB, IEC, or REB, as applicable, and an executed data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Groups:
- Prostatic Artery Embolization (PAE) Procedure: This will be a single arm, uncontrolled, non-blinded study of Prostatic Artery Embolization (PAE) using HydroPearl Beads in a small population of subjects with benign prostate hyperplasia (BPH)
  HydroPearl® compressible microspheres: Embolic material
Period: Overall Study
Arm/Group | Prostatic Artery Embolization (PAE) Procedure
Started | 12
Completed | 10
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- PAE Procedure: This will be a single arm, uncontrolled, non-blinded study of PAE using HydroPearl Beads in a small population of subjects with benign prostate hyperplasia (BPH)
  Prostatic Artery Embolization (HydroPearl® compressible microspheres): Embolic material
Arm/Group | PAE Procedure
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in IPSS at 6 Months
Description: The International Prostate Symptom Score (IPSS) includes 7 Likert-type questions related to symptoms with scores ranging from 0 to 5, where 0 is less severe. The IPSS is a written screening tool used to: screen for, rapidly diagnose, track the symptoms of, and suggest management of the symptoms of the disease benign prostatic hyperplasia (BPH). Total scores are determined to be Mild (1-7), Moderate (8-19), or Severe (20-35).
Time Frame: baseline to 6 months following the procedure
Population: Data are reported for all participants with both baseline and Month 6 data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PAE Procedure
Number analyzed (Participants) | 11
score on a scale | -9.64 (9.04)

2. Secondary Outcome: Mean Change in Quality of Life Scores at 6 Months
Description: The QoL question of the International Prostate Symptom Score (IPSS) is a single question related to the symptoms of the disease benign prostatic hyperplasia (BPH) and ranges from 0 to 6. Lower scores indicate a higher quality of life.
Time Frame: baseline to 6 months following the procedure
Population: Data are reported for all participants with both baseline and Month 6 data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PAE Procedure
Number analyzed (Participants) | 11
score on a scale | -2.00 (1.41)

3. Secondary Outcome: Mean Change in Urine Flow
Description: Urine flow will be measured to determine the maximum rate of urine flow (Qmax), which is measured in mL per second (mL/s)
Time Frame: Baseline to 6 months following the procedure
Measure: Mean (Standard Deviation); unit: mL/s
Arm/Group | PAE Procedure
Number analyzed (Participants) | 10
mL/s | 0.26 (5.25)

4. Secondary Outcome: Mean Change in Prostate Volume
Description: Change in the prostate size measured in grams (g).
Time Frame: baseline to 6 months following the procedure
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | PAE Procedure
Number analyzed (Participants) | 10
grams | -21.10 (24.63)

5. Secondary Outcome: Mean Percent of Prostate Infarcted
Description: Individual percentage of prostate infarcted determined using manual demarcation of non-enhancing areas within the prostate on serial axial slices of post contrast MRI images and data aggregated for the group to report mean percent.
Time Frame: 6 months following the procedure
Measure: Mean (Standard Deviation); unit: percent entire prostate volume infarcted
Arm/Group | PAE Procedure
Number analyzed (Participants) | 10
percent entire prostate volume infarcted | 23 (9.19)

6. Secondary Outcome: Incidence of Treatment Related Adverse Events (Proportion)
Description: Proportion of participants that experience adverse events considered related to the PAE procedure.
Time Frame: up to 3 months following the procedure
Measure: Number; unit: proportion of participants
Arm/Group | PAE Procedure
Number analyzed (Participants) | 12
proportion of participants | 0.83

7. Secondary Outcome: Incidence of Treatment Related Adverse Events (Percent)
Description: Percent of participants that experience adverse events considered related to the PAE procedure.
Time Frame: up to 3 months following the procedure
Measure: Number; unit: percentage of participants
Arm/Group | PAE Procedure
Number analyzed (Participants) | 12
percentage of participants | 83.3

ADVERSE EVENTS:
Time Frame: From the time of the PAE procedure through 12-Month Follow-Up.
Arm/Group | PAE Procedure
All-Cause Mortality (participants affected / at risk) | 1/12
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PAE Procedure (N=12)
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1)
Failure to Thrive (General disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PAE Procedure (N=12)
Dysuria (Renal and urinary disorders) | 5 (5)
Erectile Dysfunction (Reproductive system and breast disorders) | 2 (2)
Exacerbation of Hypertension (Cardiac disorders) | 1 (1)
Heaviness in distal left penis (Injury, poisoning and procedural complications) | 1 (1)
Heaviness in left lower buttock (Musculoskeletal and connective tissue disorders) | 1 (1)
Intermittency (Renal and urinary disorders) | 1 (1)
Heat sensation in pelvic area (Musculoskeletal and connective tissue disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Rectal bleeding (Gastrointestinal disorders) | 2 (2)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Strong urinary smell (Infections and infestations) | 1 (1)
Strong yellow urine color (Infections and infestations) | 1 (1)
Urgency (Renal and urinary disorders) | 1 (1)
Retrograde ejaculation (Reproductive system and breast disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Straining (Renal and urinary disorders) | 1 (1)
Pain in Groin (Post Embolization Syndrome) (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (Post Embolization Syndrome) (General disorders) | 1 (1)
Blotches on Penis (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT04398966/Prot_SAP_000.pdf